CLINICAL TRIAL: NCT01421797
Title: Evaluation of Adrenal Androgens in Normal and Obese Girls After Suppression and Stimulation (JCM022)
Brief Title: Evaluation of Adrenal Androgens in Normal and Obese Girls After Suppression and Stimulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Virginia (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of California, San Diego (Other)
Responsible Party: Principal Investigator, Christine Burt Solorzano, Assistant Professor of Pediatrics, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 12702; JCM022 (Other: University of Virginia); U54HD028934-18 (NIH); 12702 (Other: University of Virginia Institutional Review Board for Health Sciences Research)
Record Dates: First submitted 2011-08-19; First posted 2011-08-23 (Estimated); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Hyperandrogenemia; Polycystic Ovary Syndrome; Obesity
MeSH Terms: conditions — Polycystic Ovary Syndrome; Obesity | interventions — Dexamethasone; Cosyntropin; Adrenocorticotropic Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dexamethasone, Cortrosyn (Experimental): Dexamethasone given 1 mg PO Cortrosyn given single IV bolus 0f 0.25 mg
  Interventions: Drug: Dexamethasone; Drug: Cortrosyn

INTERVENTIONS:
Drug: Dexamethasone — 1 mg PO
Drug: Cortrosyn — single IV bolus of 0.25 mg will be administered
  Other Names: ACTH

SUMMARY:
Women with polycystic ovary syndrome (PCOS) often have irregular menstrual periods, too much facial and body hair, and weight gain. Women with PCOS also have a hard time becoming pregnant. Girls with high levels of the male hormone testosterone often develop PCOS as adults. Some girls with high levels of male hormone will develop normal hormone levels as they grow up, but most girls continue to have high levels of male hormone as adults. The purpose of this study is to understand where the male and female hormones come from in girls as they get older. The investigators think the adrenal gland, makes most of the hormones in young girls and that the ovary and the adrenal gland make these hormones in older girls. The investigators would like to find out whether an overactive adrenal gland makes these hormones higher in girls who are overweight, compared to those who are not overweight.

DETAILED DESCRIPTION:
We propose that the adrenal gland is the predominant source of the early morning rise in progesterone and testosterone which is more marked in early puberty. Specifically, we hypothesize that dexamethasone administration at 22:00 will be associated with a dampened progesterone and testosterone rise the subsequent morning in normal girls. We also propose that the adrenal gland is the source of the excess androgen production in young obese girls, and that dexamethasone will decrease their early morning testosterone and progesterone levels. We will explore the hypothesis that functional adrenal hyperandrogenism, or ACTH hyperresponsiveness, is one mechanism underlying this excess adrenal androgen production seen in obesity.

ELIGIBILITY:
Inclusion Criteria:

* Normal and obese (>95th BMI%) females
* Weight of 24 kg or more
* Early to late puberty (expected age range 7-18)
* Screening labs within age-appropriate normal range, with the exception of a mildly low hematocrit (see below) and the hormonal abnormalities inherent in obesity which could include mildly elevated LH, lipids, testosterone, prolactin, DHEAS, E2, glucose, and insulin; and decreased follicle-stimulating hormone (FSH) and/or sex hormone-binding globulin (SHBG)

Exclusion Criteria:

* Screening labs outside of age-appropriate normal range
* Hemoglobin <12 mg/dL and hematocrit<36% (Subjects will be offered the opportunity to take iron supplementation for 60 days if their hematocrit is slightly low (33-36%) (suggestive of iron deficiency anemia) and will then return for retesting of their hemoglobin/hematocrit. If still <36%, they will be excluded.)
* Morning Cortisol <5 g/dL
* 17-hydroxyprogesterone >295 ng/dL
* Weight<24 kg
* History of Cushing's syndrome or adrenal insufficiency
* Pregnant (self reported)

Ages: 7 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 84 (Estimated)
Dates: Start 2006-10-10 (Actual); Primary Completion 2024-08-27 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in progesterone concentrations from the 2100-2300 time block to the 0500-0700 time block in normal weight girls compared to overweight girls. | Time frame for the study will be 14 hours (Sampling begins at 1900 hrs and proceeds through 0800 hours the following morning).
  A primary endpoint for analysis in this study is the change in progesterone concentrations from the 2100-2300 time block to the 0500-0700 time block in normal weight girls compared to overweight girls.

SECONDARY OUTCOMES:
Overnight changes in male and female hormones in response to ACTH suppression | 14 hours (Sampling begins at 1900 hours and proceeds through 0800 the following morning)
  Secondary endpoints will include overnight changes in testosterone, estradiol, cortisol, dehydroepiandrosterone (DHEA), and luteinizing hormone (LH) pulse patterns in response to adrenocorticotropic hormone (ACTH) suppression. These secondary endpoints will be evaluated in a similar manner to the primary endpoint.
Response to ACTH stimulation in normal weight and overweight girls | 14 hours (1900 - 0800 hrs)
  Examine the differences in hormone responses to ACTH in normal weight and overweight girls.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Burt Solorzano, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Center for Research in Reproduction, Charlottesville, Virginia, United States